CLINICAL TRIAL: NCT04727580
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-group Clinical Trial to Study the Efficacy and Safety of HSK7653 in Chinese Patients with Impaired Glucose Tolerance
Brief Title: HSK7653 in Chinese Patients with Impaired Glucose Tolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK7653-202
Record Dates: First submitted 2021-01-21; First posted 2021-01-27 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Impaired Glucose Tolerance
Keywords: Impaired Glucose Tolerance; DPP-4 inhibitor; Prediabetes
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HSK7653 10 mg (Experimental)
  Interventions: Drug: HSK7653 10mg Q2W
- HSK7653 25 mg (Experimental)
  Interventions: Drug: HSK7653 25mg Q2W
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK7653 10mg Q2W — HSK7653 5mg (2 tablets) and placebo of HSK7653 25mg (1 tablet) Q2W, oral, Day1 to week12
  Arms: HSK7653 10 mg
Drug: HSK7653 25mg Q2W — HSK7653 25mg (1 tablet) and placebo of HSK7653 5mg (2 tablets) Q2W, oral, Day1 to week12
  Arms: HSK7653 25 mg
Drug: Placebo — Placebo of HSK7653 25mg (1 tablet) and placebo of HSK7653 5mg (2 tablets) Q2W, oral, Day1 to week12
  Arms: Placebo

SUMMARY:
This study is being done to evaluate the efficacy, safety of HSK7653 in chinese participants with impaired glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance;
* BMI (Body Mass Index) in the range of ≥ 18.0 kg/m2 to ≤ 35.0 kg/m2 at screening;

Exclusion Criteria:

* History of diabetes mellitus;
* History of severe endocrine disease, uncured cancer, acute pancreatitis prior to informed consent;
* Current uncontrolled hypertension, serious nephropathy prior to informed consent;
* Serious Heart Failure (class III-IV of the New York Heart Association functional classification), serious Arrhythmia, and Stroke within 6 months prior to informed consent;
* Serious gastrointestinal disease within 2 weeks prior to informed consent;
* Serious infection, trauma, and surgery within 3 months prior to informed consent;
* History of treatment with Glucagon-like peptide 1(GLP-1) analogues, Dipeptidyl-Peptidase 4(DPP-IV) inhibitor;
* Treatment with drugs that affect glucose metabolism within 8 weeks prior to informed consent;
* Hemoglobin (HGB) < 10.0 g/dL(100 g/L);
* Alcohol abuse within 6 months or drug abuse history within 5 years prior to informed consent;
* Active infectious diseases;
* Participation in another trial with an investigational drug or instrument within 3 months prior to informed consent;
* Women who are nursing or pregnant, or subjects with birth plans;
* Other protocol-defined inclusion/exclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Plasma Glucose AUC 0-3h for Meal Tolerance Test (MTT) at Week 12 | Baseline and Week 12
  Plasma glucose AUC 0-3 hours for MTT was measured at Baseline (Week 0) and at Week 12. After fasting for ≥8 hours, blood samples for glucose measurement were drawn at 0 minutes (at standard meal loading), 30 minutes, 60 minutes, 90 minutes, 120 minutes, and 180 minutes. At Week 12, participants received study drug or placebo 50 minutes prior to consuming a standard meal.

SECONDARY OUTCOMES:
Change From Baseline in Insulin AUC 0-3h for Meal Tolerance Test (MTT) at Week 12 | Baseline and Week 12
Change From Baseline in C-peptide AUC 0-3h for Meal Tolerance Test (MTT) at Week 12 | Baseline and Week 12
Change From Baseline in Fasting Glucose at Week 12 | Baseline and Week 12
Change From Baseline in Fasting Insulin at Week 12 | Baseline and Week 12
Change From Baseline in Fasting C-peptide at Week 12 | Baseline and Week 12
Change From Baseline in HOMA-IS at Week 12 | Baseline and Week 12
Change From Baseline in HOMA-β at Week 12 | Baseline and Week 12
Change From Baseline in Hemoglobin A1c (HbA1c) at Week 12 | Baseline and Week 12
Change From Baseline in Plasma Glucose Area Under the Curve 0 to 3 Hours (AUC 0-3 Hrs) for Oral Glucose Tolerance Test (OGTT) at Week 10 | Baseline and Week 10
Incidence of Treatment-Emergent Adverse Events | Baseline and Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No